CLINICAL TRIAL: NCT03150004
Title: A Phase II Study of the Efficacy and Pharmacogenomics of Cladribine-based Salvage Chemotherapy in Patients with Relapse/Refractory and Secondary Acute Myeloid Leukemia (AML) and High Risk Myelodysplastic Syndrome (MDS)
Brief Title: Efficacy and Pharmacogenomics of Cladribine Based Salvage Chemotherapy in Patients with Relapse/Refractory and Secondary Acute Myeloid Leukemia (AML) and High Risk Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No longer have funding support to complete the pharmacogenetics component.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Ehab L Atallah, Professor, Department of Medicine, Division of Hematology/Oncology, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO29327
Record Dates: First submitted 2017-05-02; First posted 2017-05-11 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: Acute myeloid leukemia; AML; salvage chemotherapy; CLAG-M; relapse acute myeloid leukemia; secondary acute myeloid leukemia; phase II; pharmacogenomics; myelodysplastic syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Cladribine; Cytarabine; Mitoxantrone; Granulocyte Colony-Stimulating Factor; Clinical Protocols; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CLAG-M regimen (Experimental): Subject's treatment cycle is 30 days.
  Interventions: Drug: Cladribine, Cytarabine, Mitoxantrone, G-CSF (CLAG-M) regimen
- CLLDAC regimen (Experimental): Subject's treatment cycle is 30 days. Subject may be treated on an outpatient basis (CLLDAC arm only). In addition, subjects who fail to achieve a CR/CRi after the first 30-day cycle may receive a second cycle of CLLDAC, per the discretion of the treating physician. Subjects who receive this second cycle should begin cycle 2 no later than 49 days after cycle 1.
  Interventions: Drug: Cladribine and Cytarabine (CLLDAC) Regimen

INTERVENTIONS:
Drug: Cladribine, Cytarabine, Mitoxantrone, G-CSF (CLAG-M) regimen — Subjects will be started on CLAG-M regimen, which consists of the following:
  * Cladribine 5 mg/m^2 IV over two hours on days 1-5;
  * Cytarabine 2 gm/m^2 IV over four hours on days 1-5
  * Mitoxantrone 10 mg/m^2 IV on days 1-3;
  * G-CSF at a dose of 300 μg on days 0-5.
  Other Names: Leustatin; AraC; Cytosar; Novantrone; filgastim; Neupogen; Granix; Zarxio
  Arms: CLAG-M regimen
Drug: Cladribine and Cytarabine (CLLDAC) Regimen — * Cladribine 5 mg/m^2 IV over two hours on days 1-5;
  * Cytarabine 20 mg/m^2 subcutaneous injection on days 1-10;
  Other Names: Leustatin; Cytosar
  Arms: CLLDAC regimen

SUMMARY:
This is a prospective phase II clinical study planned to be conducted at the Medical College of Wisconsin (MCW). After meeting the study criteria and enrollment, patients will be treated with a cladribine based salvage regimen and followed at periodic intervals to determine the primary and secondary objectives.

DETAILED DESCRIPTION:
STUDY RATIONALE:

The optimal treatment regimen for relapsed/refractory AML and high risk MDS progressing after hypomethylating agents is unknown. Although several chemotherapy options are available, there is no universally accepted regimen to date. Cladribine based salvage regimens have been frequently used at the investigators' center. However, it is uncertain to predict which patients are likely to respond to cladribine-based salvage or experience treatment-related toxicities. While studies have demonstrated that achievement of MRD negative complete remission (CR) is likely to be associated with a better overall survival (OS), there is limited prospective data evaluating the role of minimal residual disease (MRD) in the setting of relapsed/refractory disease. Through this study, the investigators aim to demonstrate the influence of achieving MRD negative CR on survival of patients with relapsed/refractory AML/high risk MDS treated with cladribine-based salvage therapy. In addition to the conventionally used predictive factors, we aim to incorporate pharmacogenomics to assess the efficacy and toxicity of therapy.

PRIMARY OBJECTIVE:

To determine the CR rate and achievement of MRD negativity after treatment with Cladribine based salvage chemotherapy regimen in patients with relapse/refractory AML/high risk MDS.

SECONDARY OBJECTIVES:

1. To determine the progression free survival (PFS) and overall survival (OS) of patients treated with a cladribine based salvage chemotherapy regimen.
2. To study the pharmacogenomics of patients receiving a cladribine based salvage and determine its influence on survival, CR rate and MRD negativity.
3. Determination of disease- or patient-related factors that predict MRD negativity and survival with a cladribine based salvage regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of informed consent.
2. Morphologically documented:

   * Primary Acute Myeloid Leukemia (AML) or
   * AML secondary to Myelodysplastic Syndrome (MDS) or myeloproliferative neoplasm (MPN), or
   * Therapy related AML (t-AML), as defined by World Health Organization (WHO) criteria.
   * Subjects with high risk MDS after failure of hypomethylating agents are also eligible.
3. Subjects must meet one of the following criteria:

   * In first or subsequent relapse or refractory status, with or without prior hematopoietic stem cell transplant (HSCT) OR
   * Subjects with MDS or MPN transformed to AML will be eligible even if they had not received prior therapy for AML.
   * Subjects with high risk MDS after failure of hypomethylating agents.
4. Eastern Cooperative Oncology Group (ECOG) performance score 0-3.
5. It is not known what effects this treatment has on human pregnancy or development of the embryo or fetus. Therefore, female subjects participating in this study should avoid becoming pregnant, and male subjects should avoid impregnating a female partner. Non- sterilized female subjects of reproductive age and male subjects should use effective methods of contraception through defined periods during and after study treatment as specified below.

   Female subjects must meet one of the following:
   * Postmenopausal for at least one year before the screening visit, or
   * Surgically sterile, or if they are of childbearing potential, agree to practice two effective methods of contraception from the time of signing of the informed consent form through 90 days after the last dose of study drug, AND
   * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, or
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)

   Male subjects, even if surgically sterilized (i.e., status post vasectomy), must agree to one of the following:
   * Practice effective barrier contraception during the entire study treatment period and through 90 days after the last study drug dose, OR
   * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
6. Ability to understand a written informed consent document and the willingness to sign it.
7. Subjects must meet the following clinical laboratory criteria:

CLAG-M Arm Only:

For abnormalities in liver function tests, elevation thought to be due to hepatic infiltration by AML, Gilbert's syndrome or hemolysis would not be treated as exclusion criteria.

* Absolute neutrophil count ≥1,000/mm^3 Unless related to AML
* Platelets ≥75,000/mm^3 Unless related to AML
* Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN) (if elevated, then complete direct bilirubin).
* AST(SGOT)/ALT Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN
* Creatinine clearance ≥ 30 mL/min
* Resting left ventricular ejection fraction ≥ 45%

CLLDAC ARM ONLY:

* Absolute neutrophil count ≥ 1,000/mm^3 unless related to AML
* Platelets ≥ 75,000/mm^3 unless related to AML

Exclusion Criteria:

1. Acute Promyelocytic Leukemia.
2. Active infection not well controlled by antibacterial or antiviral therapy.
3. Pregnant or breast feeding women.
4. Participation in clinical trials with other investigational agents not included in this trial, throughout the duration of this trial. Participation of follow-up portion of another clinical trial will not exclude patient from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
CLAG-M Arm: Minimal residual disease (MRD) complete remission (CR) | Day 35
  The number of participants who achieve MRD CR (see Cheson 2003, Cheson 2006 in the references below).
CLLDAC Arm: Minimal residual disease (MRD) complete remission (CR) | Day 35
  The number of participants who achieve MRD CR following one cycle of therapy (see Cheson 2003, Cheson 2006 in the references below).
CLLDAC Arm: Subjects receiving a second cycle. | Day 70
  The number of subjects who require a second cycle of CLLDAC.
Overall survival | Year 4
  The number of participants still alive following CLAG-M chemotherapy.
Progression-free survival | Year 4
  The number of participants who don't experience progressive disease.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Atallah, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheson BD, Greenberg PL, Bennett JM, Lowenberg B, Wijermans PW, Nimer SD, Pinto A, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Gore SD, Schiffer CA, Kantarjian H. Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia. Blood. 2006 Jul 15;108(2):419-25. doi: 10.1182/blood-2005-10-4149. Epub 2006 Apr 11. PMID 16609072
- [Background] Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, Schiffer CA, Doehner H, Tallman MS, Lister TA, Lo-Coco F, Willemze R, Biondi A, Hiddemann W, Larson RA, Lowenberg B, Sanz MA, Head DR, Ohno R, Bloomfield CD; International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol. 2003 Dec 15;21(24):4642-9. doi: 10.1200/JCO.2003.04.036. PMID 14673054